CLINICAL TRIAL: NCT04535648
Title: Rapid Identification and Clinical Transformation of Various Enterovirus Genotypes Based on CRISPR Technology
Brief Title: Detection of Enterovirus Genotypes by CRISPR Technology
Status: Withdrawn | Type: Observational
Why Stopped: This clinical trial has been terminated。
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: EV-CRISPR.001
Record Dates: First submitted 2020-08-25; First posted 2020-09-02 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Enterovirus Infections
MeSH Terms: conditions — Enterovirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Samples of feces, blood and cerebrospinal fluid (the remainder of routine testing samples) from 500 children with suspected or confirmed enterovirus infection were collected for detection by the CRISPR technique.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non-invasive detection method: CRISPR techonology — This study was a laboratory diagnostic study without any intervention.
  Other Names: No intervention

SUMMARY:
CRISPR-enterovirus detection system was constructed in this study for detection variety genotypes of enterovirus rapidly in children suspected or diagnosed as enterovirus infection.

DETAILED DESCRIPTION:
To construct CRISPR-enterovirus detection system, we screened the targets, primers and CrRNA and evaluated the capability of this detecting system. Samples of feces, blood and cerebrospinal fluid (the remainder of routine testing samples) from 500 children with suspected or confirmed enterovirus infection were examined using the CRISPR technique. To evaluate the CRISPR-enterovirus detection system, real-time PCR and traditional PCR as comparison method was implemented. The method of real-time PCR and traditional PCR were used to detect enterovirus and analyze the genotypes of enterovirus, respectively. According to the results of CRISPR-enterovirus detection system and the comparison method, the positive coincidence rate, negative coincidence rate and consistency of the two methods were calculated. Furthermore, the sensitivity and specificity of the CRISPR-enterovirus detection system for detection of enterovirus were calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically suspected or confirmed enterovirus infection

Exclusion Criteria:

* Patients with clinical diagnosis of non-enterovirus infection

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who came to the Children's Hospital of Fudan University and were diagnosed with enterovirus infection.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Successful construction of CRISPR-enterovirus detection system | At enrollment
  It is a binary variable ("yes/no").If the system meet all the following criteria, it would be setted into "yes" .According to the results of CRISPR-enterovirus detection system and the comparison method：
  1. the positive coincidence rate and negative coincidence rate are both over 95.0%;
  2. the value of Kappa using to express the consistency of those two methods is over 0.75;
  3. the sensitivity and specificity of the CRISPR-enterovirus detection system for detection of enterovirus are over 90.0% and 95.0%;
  4. the coefficient of variation between batches is less 15.0%, and each batch detection takes less than 1 hour.

CONTACTS AND LOCATIONS:
Overall Officials: Liling Qian, Study Director — Children's Hospital of Fudan University

IPD SHARING:
Plan to Share IPD: No